CLINICAL TRIAL: NCT06541366
Title: Physical Capacity of Spina Bifida and Factors Affecting During Pregnancy: A Case Control Study
Brief Title: Physical Capacity of Spina Bifida and Factors Affecting
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammed ARCA, Dr., Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: SBUGaziYasargil21
Record Dates: First submitted 2024-07-14; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism | interventions — Case-Control Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: The case group consisted of patients who were diagnosed in the Neonatal Intensive Care Unit (39 children), and who applied to the Physiotherapy and Rehabilitation Department from the centers outside for physiotherapy needs (9 children).
  Interventions: Other: case-control study
- Control: the children who were at the same age group between the same dates, did not have any diseases related to the neuromuscular system, and hospitalized for any other reason.
  Interventions: Other: case-control study

INTERVENTIONS:
Other: case-control study — physical examination and Survey Form

SUMMARY:
Objective: It was aimed to evaluate the physical characteristics of the cases with spina bifida and to review the factors that may affect the etiology of the disease.

Methods: 48 cases with spina bifida and 48 control groups in other disease groups evaluated. A physiotherapist physically evaluated the cases after their personal information was obtained. A survey form examining the possible factors in the etiology of spina bifida was applied to the families.

DETAILED DESCRIPTION:
The study was carried out with the participation of 48 cases with spina bifida between the ages of 0 and 2 evaluated in XXXXXX Training and Research Hospital (XXXXX) Pediatric Clinics and 48 control groups in other disease groups in response to each case.

The case group consisted of patients who were diagnosed in the Neonatal Intensive Care Unit between February 2019 and January 2020 (39 children), and who applied to the Physiotherapy and Rehabilitation Department from the centers outside for physiotherapy needs (9 children).

ELIGIBILITY:
Inclusion Criteria:

* spina bifida between the ages of 0 and 2

Exclusion Criteria:

* control group was formed through random selection among the children who were at the same age group between the same dates, did not have any diseases related to the neuromuscular system, and hospitalized for any other reason.

Ages: 0 Years to 2 Years | Sex: All
Age Groups: Child
Study Population: The case group consisted of patients who were diagnosed in the Neonatal Intensive Care Unit between February 2019 and January 2020 (39 children), and who applied to the Physiotherapy and Rehabilitation Department from the centers outside for physiotherapy needs (9 children). The control group was formed through random selection among the children who were at the same age group between the same dates, did not have any diseases related to the neuromuscular system, and hospitalized for any other reason.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Results of Groups | 1-2 month
  FACTORS AFFECTING DURING PREGNANCY QUESTIONARRE
Antropomethric measures | 1-2 month
  body mass index (kg/cm2)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Diyarbakır Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No